CLINICAL TRIAL: NCT01617850
Title: Efficacy of Physical Exercise in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Mette Krintel Petersen, assistant professor,PT, Ph.D, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20100297
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Heart Disease; Heart Failure; Ischemic Heart Diseases
MeSH Terms: conditions — Coronary Disease; Heart Failure; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- optimized physical exercise training (Experimental): Intervention: Supervised physical exercise training x3 weekly for 12 weeks
  Interventions: Other: Supervised physical exercise training x3 weekly for 12 weeks
- conventional group (Active Comparator): Intervention: Supervised physical exercise training x2 weekly for 8 weeks
  Interventions: Other: Supervised physical exercise training x2 weekly for 8 weeks

INTERVENTIONS:
Other: Supervised physical exercise training x3 weekly for 12 weeks — Physical exercise training 1 hour per session. The exercise rehabilitation programme is carried out as group training with individual supervision. At each exercise session two experienced physiotherapist are leading the physical exercise training. Standardized physical exercise guidelines for each training session is described and followed. It consists of the following interventions: Warm up, aerobe fitness, muscle strength training and individual education and instruction in life stills changes in relation to physical activity.
  Arms: optimized physical exercise training
Other: Supervised physical exercise training x2 weekly for 8 weeks — Physical exercise training is carried out for 1 hour per session. The exercise rehabilitation programme is carried out as group training with individual supervision. At each exercise session two-experienced physiotherapist are leading the physical exercise training. Standardized physical exercise guidelines for each training session is described and followed. It consists of the following interventions: Warm up, aerobe fitness, muscle strength training and individual education and instruction in life stills changes in relation to physical activity.
  Arms: conventional group

SUMMARY:
Physical rehabilitation is a key element in the treatment of patients with cardiovascular diseases, and recent evidence has shown that supervised exercise programmes can prevent cardiovascular events, improve physical function and quality of life. Individualized exercise prescription based on appropriate frequency, intensity and duration is recommended. Furthermore, recent studies have shown that physical cardiac exercise training can influence inflammation of the vessel wall and hence reduce development of arteriosclerosis in coronary vessels. In the literature are divergent conclusions on appropriate frequency and duration of physical rehabilitation programs in order to improve physical function and reduce arteriosclerosis.

The purpose of this study is to investigate the efficacy of an optimized physical rehabilitation programme compared to a conventional programme on physical fitness, health related quality of life and vascular inflammation.

DETAILED DESCRIPTION:
Both trial groups carry out physical exercise training in groups. The exercise training is instructed by two physiotherapists with expertise in cardiac rehabilitation. Each training session takes 60 minutes and is based on current evidence for physical training for IHD and CHF patients. Exercise intensity progresses within the first week of the training program from moderate intensity (40-59% of VO2max), to high intensity (60-84% of VO2max). Exercise intensity of the individual training sessions is monitored by heart rate.

The training program includes the following:

Warm-up and stretching: Each training sessions starts 10 min. warm-up and ends with 5 min. stretching.

Aerobic exercise : Takes place on treadmill, stairs, ergometer bikes and interval training with different strength-endurance exercises.

Muscle strength: Is performed on machines with weight training equipment or by floor exercises. 10-15 repetitions are performed with a load equivalent to 50-60% of 1 RM.

The exercise programs for both groups are performed using a standardized exercise protocol.

All patients per a sub-maximal and a maximal exercise test prior to participation in the physical exercise training program.

ELIGIBILITY:
Inclusion Criteria:

Patients prescribed to physical exercise training at Skejby University Hospital with:

* stable and unstable angina pectoris,
* acute myocardial infarction with and without ECG changes
* chronic heart failure

Exclusion Criteria:

* patients with BMI>35
* patients with musculoskeletal or neurological diseases that unable them to participate in physical exercise training programmes
* patients who can not read or understand danish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity measured as maximal oxygen uptake (V02 max) | Changes in aerobic capacity between baseline and end of intervention (8 respectively 12 weeks). Follow-up data 6 and 12 month after end of intervention
  Cardiopulmonary exercise testing (CPX) using breath by breath gas-analysis measures variables related to cardiorespiratory function, including expiratory ventilation and pulmonary gas exchange (oxygen uptake (VO2) and carbon dioxide (VCO2). Along with the ECG, heart rate and blood pressure these measures allows for quantitatively linking metabolic, cardiovascular and pulmonary responses to exercise. The standard expression of aerobic working capacity is the maximum VO2.
  VO2 max reached during a symptom-limited incremental CPX protocol is commonly expressed as O2 per kg-1 per min -1.

SECONDARY OUTCOMES:
Muscle strength | Changes from baseline in muscle strength at end of intervention (8 respectively 12 weeks)
  Isometric muscle strength and muscle power are essential determinants for physical performance. Maximal isometric muscle strength is defined as a maximal volunteer contraction at a specific range of motion, and muscle power as the ability to produce high force rapidly.
  Isometric volunteer knee extension is measured with the patients sitting in a adjustable dynamometer chair (Good Muscle Strength, Metittur®) and measurement of leg extensor power is measured using a Nottingham Power Rig ®
VCAM-1 | Changes in VCAM-1(pg/ml) between baseline and end of intervention (8 respectively 12 weeks). Follow-up 6 and 12 month after end of intervention.
  VCAM-1 is an endothelial cell protein, which is gate, when leukocytes reside on the intima of the vessel wall. TNF-alpha stimulates endothelial cell to membrane expression of VCAM-1, where leukocytes can adhere to endothelial cell s and influence inflammation of the vessel wall. VCAM-1 is thus a specific inflammation marker in the vessel wall, and hence development of arteriosclerosis in coronary vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Christian Djuurhuus, professor,MD, Study Chair — Institute of Clinical Medicine, Aarhus University, Department of Physio- and Occupationaltherapy, Aarhus University Hospital, Skejby
Locations (1):
- Department of Physiotherapy and Occupational therapy, Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark